CLINICAL TRIAL: NCT06194461
Title: A LOng-term Follow-up Master Protocol for Participants Who Received Cell or Gene Therapies in Other AstraZeneca StUdieS (LOCUS)
Brief Title: LTFU for All Cell and Gene Therapy Studies
Acronym: LOCUS
Status: Not yet recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9341C00001
Record Dates: First submitted 2023-12-07; First posted 2024-01-08 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma; Prostate Cancer
Keywords: Cell Therapy; Gene Therapy; Long term follow up; LTFU; Hepatocellular carcinoma; Prostate cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AZD5851: Follow-up for up to 15 years of subjects who received AZD5851 in study NCT06084884
  Interventions: Biological: AZD5851
- AZD0754: Follow-up for up to 15 years of subjects who received AZD0754 in study NCT06267729
  Interventions: Biological: AZD0754

INTERVENTIONS:
Biological: AZD5851 — Safety follow-up for up to 15 years of subjects who received AZD5851 in study NCT06084884.
  Groups: AZD5851
Biological: AZD0754 — Safety follow-up for up to 15 years of subjects who received AZD0754 in study NCT06267729.
  Groups: AZD0754

SUMMARY:
Master LTFU study will monitor the long-term safety and tolerability of cell or gene therapy study participants from AstraZeneca for up to 15 years post last cell or gene therapy treatment.

DETAILED DESCRIPTION:
This is a multi-centre and multinational basket study that will monitor the long-term safety and tolerability of cell or gene therapies in participants that have taken part in other AstraZeneca cell or gene therapy studies for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

1. The participant has received a cell or gene therapy in another AstraZeneca protocol.
2. Provision of signed and dated, written informed consent before any study-specific procedures.

Exclusion Criteria:

Not applicable

-

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have been treated with Cell/Gene therapy products in AstraZeneca clinical trials.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-09-17 (Estimated); Primary Completion 2041-11-29 (Estimated); Study Completion 2041-11-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of specific AEs | Maximum of 15 years post dosing
  To determine long-term safety of previous treatment with applicable cell and gene therapy products

SECONDARY OUTCOMES:
Disease progression status and Overall survival | Maximum of 15 years post dosing.
  To determine long-term efficacy follow-up after previous treatment with a cell or gene therapy product
Kinetics parameters that indicate persistence (eg, Clast and Tlast) | Maximum of 15 years post dosing
  To characterise the long-term persistence of the cell or gene therapy product.

CONTACTS AND LOCATIONS:
Locations (23):
- United States (18):
  - Research Site, Phoenix, Arizona
  - Research Site, Duarte, California
  - Research Site, Orange, California
  - Research Site, San Francisco, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Jacksonville, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Westwood, Kansas
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Hackensack, New Jersey
  - Research Site, New York, New York
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Houston, Texas
- Research Site, East Melbourne, Australia
- Japan (3):
  - Research Site, Kashiwa
  - Research Site, Kyoto
  - Research Site, Osakasayama-shi
- Research Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal
  Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/